CLINICAL TRIAL: NCT05774145
Title: Dexmeditomedine Versus No Sedation in Management of Agitation in COPD Patients Receiving Noninvasive Ventilation
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Hoda sultan, Principle investigator, Assiut University
Other Study IDs: Dexmeditomedine Versus No Seda
Record Dates: First submitted 2023-02-22; First posted 2023-03-17 (Actual); Last update posted 2023-03-17 (Actual); Status verified 2023-03

CONDITIONS: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim is to compare sedation using dexmedetomidine to sedation -free approach in management of agitated COPD patients receiving NIV

DETAILED DESCRIPTION:
The aim is to compare sedation using dexmedetomidine to sedation -free approach in management of agitated COPD patients receiving NIV

ELIGIBILITY:
Inclusion critera

* age>18
* Agitation
* NIV intolerance Exclusion criteria
* cardiac dysfunction
* Hepatic dysfunction
* Haemodynamic instability

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: observational study
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2023-03 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
precedex on COPD irritable on non invasive machine | 3/2023_3/2025
  control of Agitation by RASS